CLINICAL TRIAL: NCT01636232
Title: Vitamin D Levels and Risk of Infection, Assessment for Disease Severity, and Predictor of Mortality in the Chinese Intensive Care Units: a Prospective Cohort Study
Brief Title: Vitamin D and Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Longxiang Su, Dr., Chinese PLA General Hospital
Other Study IDs: CPLAGH-2012026
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Systemic Inflammatory Response Syndrome; Sepsis
Keywords: Vitamin D; infection; disease severity; mortality; critically ill; sepsis
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Sepsis; Infections; Critical Illness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- ICU sepsis group: The ICU sepsis group consisting of 105 critically-ill cases diagnosed with sepsis upon admission and sampled within the first 24h of their ICU stay.
- ICU control group: the ICU control group including 51 critically-ill cases in whom sepsis was clinically excluded and from whom samples were taken upon admission.
- healthy control group: the healthy control group composed of 50 healthy control outpatients. For the healthy control outpatients, possibilities of acute or past chronic diseases were excluded. Moreover, we made sure that the healthy control subjects had not been hospitalized or taken vitamin-based substitutive drugs in the last 12 months, and proved normal in physical checkups and lab examinations.

SUMMARY:
The higher rate of vitamin D deficiency is spotted among patients being hospitalized or in critical condition. Especially, vitamin D level below normal prolongs hospital stay and increases incidence of adverse prognosis and pushing up mortality of a number of diseases. However, it is remain unclear the relationship between vitamin D levels and critically ill, especially infection or sepsis. In this study, the investigators evaluate the significance of vitamin D for diagnosis and other relevant assessments of ICU cases, including vitamin D's relevance to sepsis, as well as its value in severity and prognosis assessment, high-performance liquid chromatography and tandem mass spectrometry was used to detect the quantification of the total 25(OH)D in serum of critically ill patients. The investigators speculate that measurement of vitamin D could be taken as an indicator for diagnosis and assessment in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 18 years old and over;
* Entered ICU;
* Fulfilled at least two criteria of systemic inflammatory response syndrome

  * core temperature higher than 38 °C or lower than 36 °C
  * respiratory rate above 20/min, or PCO2 below 32 mmHg
  * pulse rate above 90/min, and
  * white blood cell count greater than 12,000/μl or lower than < 4,000/μl or less than 10% of bands.

Exclusion Criteria:

* patients or their relatives refused

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the subjects were selected from among inpatients who were hospitalized between October-December, 2011 in the Surgical ICU, Respiratory ICU, and Emergency ICU, Chinese PLA General Hospital.
Sampling Method: Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Patients Outcome | 28 days
  The survival time of patients more than 28 days is defined as survival. The survival time of patients less than 28 days is defined as death.
Patients Outcome | 90 days
  The survival time of patients more than 90 days is defined as survival. The survival time of patients less than 90 days is defined as death.

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Xie, MD, Study Director — Department Of Respiratory Diseases, Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

REFERENCES:
- [Derived] Su LX, Jiang ZX, Cao LC, Xiao K, Song JP, Li H, Zhang X, Yan P, Feng D, Liu CT, Li X, Xie LX. Significance of low serum vitamin D for infection risk, disease severity and mortality in critically ill patients. Chin Med J (Engl). 2013 Jul;126(14):2725-30. PMID 23876904